CLINICAL TRIAL: NCT05417412
Title: Video-visit Behavior Therapy for Anxiety and Depression in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Kaiser Permanente (Other); OCHIN, Inc. (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, V. Robin Weersing, Professor, San Diego State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R56MH125159 (NIH); R56MH125159 (NIH)
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Anxiety; Depression
Keywords: Child; Adolescent
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEP-UP (brief behavioral therapy) (Experimental): Intervention arm of open trial
  Interventions: Behavioral: Brief Behavioral Therapy

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy — 8-12 sessions of brief behavioral therapy administered by behavioral health / mental health staff at participating community health centers (CHCs)
  Other Names: STEP-UP; BBT

SUMMARY:
This project focuses on adapting and pilot testing an efficacious brief behavioral therapy (STEP-UP) for youths with anxiety or depression to be delivered as a telehealth intervention by clinic staff in low-resource community health centers (CHCs).

ELIGIBILITY:
Inclusion Criteria:

* Youth is a patient at a participating community health center (CHC) site
* Youth is clinically referred by a provider and / or has anxiety and / or depression as a diagnosis or target problem in their medical record
* Youth is in the physical and legal custody of the caretaker and is not currently involved in the foster care system
* Youth is able and willing to conduct study assessments and intervention sessions in English
* Primary caretaker is able and willing to conduct study assessments and intervention sessions in English or in Spanish
* Youth is functioning at or above the academic level of a typical 8-year-old child (i.e., placed in at least the second-grade level school across all subjects in a general education classroom)
* Primary caretaker agrees that focusing on anxiety and / or depression would be a useful primary target for treatment
* Youth has clinically significant symptoms of anxiety and / or depression by youth or caretaker report

Exclusion Criteria:

* Youth is receiving an alternate intervention for anxiety or depression
* Youth or parent reports that the youth is experiencing active suicidal ideation with plan or intent (i.e., within last three months) and / or has made a suicide attempt within the last six months
* Youth or parent reports that the youth is currently engaging in non-suicidal self-injury (i.e., within last three months)
* Youth or parent reports that the youth has experienced recent physical or sexual abuse (i.e., within last three months).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Northwest Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Youths were recruited from community health centers through electronic health record identification and clinician referral. Youth and their caregivers / guardians ("parents") were mailed letters describing the study and giving them the opportunity to opt-out of research contact. Families that did not opt-out were called by research staff, screened for initial eligibility, and consented for participation.
Groups:
- STEP-UP (Brief Behavioral Therapy): Intervention arm of open trial
  Brief Behavioral Therapy: 8-12 sessions of brief behavioral therapy administered via telehealth by behavioral health / mental health staff at participating community health centers (CHCs)
Period: Overall Study
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Started | 12 (12 youths were consented and started in treatment in the open trial)
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Youths with significant symptoms of anxiety and depression were recruited through electronic medical record screening and clinican referral. Youths were the target of treatment and the enrolled participants. As youth are minors, consent for youth participation was sought from parents, and information on youths obatined from parents / guardians in addition to youth self-report.
Groups:
- STEP-UP (Brief Behavioral Therapy): Intervention arm of open trial
  Brief Behavioral Therapy: 8-12 sessions of brief behavioral therapy administered via telehealth by behavioral health / mental health staff at participating community health centers (CHCs). Youths were the target of treatment and were the enrolled participants in the clinical trial.
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — Parent report of youth age
  Participants
    <=18 years | 12
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Parent and youth report of youth sex
  Participants
    Female | 9
    Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parent report of youth ethnicity
  Participants
    Hispanic or Latino | 4
    Not Hispanic or Latino | 8
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Parent report of youth race
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 7
    More than one race | 0
    Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants] — Data collected from targeted clinics in known geographic regions within the United States
  Participants
    United States | 12
Screen for Anxiety and Related Disorders - Parent report on child (SCARED-P) [Mean (Standard Deviation); unit: units on a scale] — Total score on the Screen for Anxiety and Related Disorders scale (parent report on youth), a dimensional measure of anxiety symptoms. Scores range from 0 to 82, and higher scores indicate greater symptom severity. Scores >= 25 may indicate the presence of an anxiety disorder.
  units on a scale | 37.17 (13.43)
Screen for Anxiety and Related Disorders - child report on self (SCARED-C) [Mean (Standard Deviation); unit: units on a scale] — Total score on the Screen for Anxiety and Related Disorders scale (youth report on self), a dimensional measure of anxiety symptoms. Scores range from 0 to 82, and higher scores indicate greater symptom severity. Scores >= 25 may indicate the presence of an anxiety disorder.
  units on a scale | 38.25 (13.24)
Mood and Feelings Questionnaire - parent report on child (MFQ-P) [Mean (Standard Deviation); unit: units on a scale] — Total score on the Mood and Feelings Questionnaire - parent report on youth (MFQ-P) a dimensional measure of depression symptoms. Scores range from 0 to 68, and higher scores indicate greater depression symptom severity.
  units on a scale | 13.25 (6.48)
Mood and Feelings Questionnaire child report on self (MFQ-C) [Mean (Standard Deviation); unit: units on a scale] — Total score on the Mood and Feelings Questionnaire - youth report on self (MFQ-C) a dimensional measure of depression symptoms. Scores range from 0 to 66, and higher scores indicate greater depression symptom severity.
  units on a scale | 21.83 (11.28)
Insurance status [Count of Participants; unit: Participants] — Parent report of family health insurance coverage
  Participants
    Private insurance | 3
    Medicaid / uninsured | 9

OUTCOME MEASURES:

1. Primary Outcome: Minimum Attendance
Description: Receipt of a minimum dose of intervention. A minimum dose was defined as 8 or more sessions of the intervention.
Time Frame: Week 16 (post-intervention)
Population: Receipt of a minimum dose of intervention was coded from electronic medical records for all 12 enrolled youths. Families who were lost to follow-up were included in these analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 12
Participants
  Attended less than 8 sessions | 5
  Attended 8 or more sessions | 7

2. Primary Outcome: Client Satisfaction Scale - Parent (CSQ-8-P)
Description: Parent ratings of satisfaction with the intervention. Ratings of "mostly" or "very" satisfied were coded as "satisfied." All other ratings were coded as "unsatisfied."
Time Frame: Week 16 (post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 12
Participants
  Satisfied | 9
  Unsatisfied | 0
  Unknown / lost to follow-up | 3

3. Primary Outcome: Client Satisfaction Scale - Child (CSQ-8-C)
Description: Youth ratings of satisfaction with the intervention. Ratings of "mostly" or "very" satisfied were coded as "satisfied." All other ratings were coded as "unsatisfied."
Time Frame: Week 16 (post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 12
Participants
  Satisfied | 10
  Unsatisfied | 0
  Unknown / lost to follow-up | 2

4. Primary Outcome: Participant Acceptability Questionnaire - Parent (PAQ-P)
Description: Parent ratings of the acceptability of the telehealth intervention. Responses were classified as "little or no technical problems" or "technical difficulties."
Time Frame: Week 16 (post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 12
Participants
  Little to no technical problems | 6
  Technical difficulties | 3
  Unknown / lost to follow up | 3

5. Primary Outcome: Participant Acceptability Questionnaire - Child (PAQ-C)
Description: Youth ratings of the acceptability of the intervention. Youths were asked whether they would recommend the intervention to a friend. Responses were included "would recommend" and "unlikely."
Time Frame: Week 16 (post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 12
Participants
  Would recommend program to a friend | 9
  Unlikely to recommend program to a friend | 1
  Unknown / lost to follow-up | 2

6. Secondary Outcome: Screen for Child Anxiety and Related Disorders - Parent (SCARED-P)
Description: Total score on the Screen for Anxiety and Related Disorders scale (parent report on youth), a dimensional measure of anxiety symptoms. Scores range from 0 to 82, and higher scores indicate greater symptom severity. Scores >= 25 may indicate the presence of an anxiety disorder.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 9
score on a scale | 30.00 (17.66)

7. Secondary Outcome: Screen for Child Anxiety and Related Disorders - Child (SCARED-C)
Description: Total score on the Screen for Anxiety and Related Disorders scale (youth report on self), a dimensional measure of anxiety symptoms. Scores range from 0 to 82, and higher scores indicate greater symptom severity. Scores >= 25 may indicate the presence of an anxiety disorder.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 10
score on a scale | 28.80 (13.66)

8. Secondary Outcome: Mood and Feelings Questionnaire - Parent (MFQ-P)
Description: Total score on the Mood and Feelings Questionnaire - parent report on youth (MFQ-P) a dimensional measure of depression symptoms. Scores range from 0 to 68, and higher scores indicate greater depression symptom severity.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 9
score on a scale | 15.22 (10.96)

9. Secondary Outcome: Mood and Feelings Questionnaire - Child (MFQ-C)
Description: Total score on the Mood and Feelings Questionnaire (youth report on self) a dimensional measure of depression symptoms. Higher scores indicate greater symptom severity. Scores range from 0 to 66, and higher scores indicate greater depression symptom severity.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 10
score on a scale | 18.00 (8.78)

10. Secondary Outcome: Symptom Impairment Scale - Parent (SIS-P)
Description: Parent rating of child impairment in school, social, and family domains from symptoms of anxiety (3 questions) and depression (3 questions). Higher scores indicate greater levels of perceived impairment. Individual questions scores range from zero (not at all impairing) to three (very much impairing), and the total score ranges from 0 to 18.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 9
score on a scale | 6.44 (4.19)

11. Secondary Outcome: Symptom Impairment Scale - Child (SIS-C)
Description: Youth self-rating of impairment in school, social, and family domains from symptoms of anxiety (3 questions) and depression (3 questions). Higher scores indicate greater levels of perceived impairment. Individual questions scores range from zero (not at all impairing) to three (very much impairing), and the total score ranges from 0 to 18.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 10
score on a scale | 7.80 (3.77)

12. Secondary Outcome: Child Avoidance Measure - Parent (CAMP)
Description: Parent rating of youth avoidance behaviors due to anxiety. Scores range from 0 to 24, and higher scores indicate greater avoidance.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 9
score on a scale | 11.78 (5.43)

13. Secondary Outcome: Child Avoidance Measure - Child (CAMP)
Description: Youth self-report rating of avoidance behaviors due to anxiety. Scores range from 0 to 24, and higher scores indicate greater avoidance.
Time Frame: Week 16 (post-intervention)
Population: Descriptive statistics at Week 16 are based on participants not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP (Brief Behavioral Therapy)
Number analyzed (Participants) | 9
score on a scale | 11.44 (5.70)

ADVERSE EVENTS:
Time Frame: Data collected from baseline (Week 0) through follow-up (Week 16)
Groups:
- STEP-UP (Brief Behavioral Therapy): Intervention arm of open trial
  Brief Behavioral Therapy: 8-12 sessions of brief behavioral therapy administered by behavioral health / mental health staff via telehealth at participating community health centers (CHCs)
Arm/Group | STEP-UP (Brief Behavioral Therapy)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
This pilot study was designed and funded prior to the COVID-19 pandemic; however, all enrollment of participants and delivery of intervention occurred after the start of the pandemic. The study was based in primary care, and the STEP-UP treatment was provided by clinical staff as part of their regular responsibilities. Results should be interpreted in this historical context of heavy demand on health care providers and facilities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT05417412/Prot_000.pdf